CLINICAL TRIAL: NCT01509781
Title: Optimal Wound Care After Simplex or Modified Radical Mastectomy With or Without Axillary Lymphadenectomy Placement of a Drain Versus the Use of Adaptive Skin Sutures; a Prospective Randomised Study
Brief Title: Suction Drain Versus the Use of Adaptive Skin Sutures After Mastectomy ± Axillary Lymphadenectomy; a Prospective Randomised Study
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute of Oncology, Hungary (Other)
Responsible Party: Principal Investigator, Dr. Zoltan Matrai, principal investigator, National Institute of Oncology, Hungary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MRM-987/2011
Record Dates: First submitted 2012-01-08; First posted 2012-01-13 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: in Situ Breast Cancer; Invasive Breast Cancer
Keywords: simple mastectomy; modified radical mastectomy; wound care; suction drain; adaptive suture
MeSH Terms: conditions — Breast Carcinoma In Situ

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Suction drain (Active Comparator): Patients in Arm A undergo simplex mastectomy or modified radical mastectomy. One plastic Redon drain (16 Ch) is placed after simplex mastectomy and two plastic Redon drains (16 Ch each) following modified radical mastectomy.
  Interventions: Procedure: Insertion of suction drain(s) following mastectomy
- Adaptive suture (Experimental): Following mastectomy, wound cavity is closed with adaptive skin sutures. No suction drain is inserted.
  Interventions: Procedure: Adaptive skin sutures.

INTERVENTIONS:
Procedure: Insertion of suction drain(s) following mastectomy — One suction drain (16 Ch Redon drain) following simple mastectomy and two following modified radical mastectomy.
  Arms: Suction drain
Procedure: Adaptive skin sutures. — Subcutis of skin flaps of the axilla and the wound edges are adapted to the chest wall and pectoralis major muscle by 8 to 24 stitches (depending on the wound surface of the breast and axilla) using 3.0 absorbable sutures, in a distance of 4-5 cm from each other in a chessboard pattern. The wound is then closed with 3.0 running subcutaneous sutures and 4.0 intracutaneous stitches. Compressive dressing is applied on the chest in the first 12-24 hours after surgery.
  Arms: Adaptive suture

SUMMARY:
The objective of this prospective randomized study is to perform qualitative and quantitative comparisons between the insertion of traditional suction drains (Arm: Suction drain) versus the application of absorbable adaptive sutures (Arm: Adaptive suture) following simplex mastectomy or modified radical mastectomy in the light of the total volume of withdrawn serum from wound cavity, the extent of early postoperative analgesic requirements and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* female patients with primary unilateral, stage 0, I or II, T3N1M0 breast cancer necessitating simple or modified radical mastectomy

Exclusion Criteria:

* age above 75 years and bad general state
* pregnancy
* autoimmune disease
* non-radical excision
* mastitis carcinomatosis
* lymphangitis carcinomatosis
* wound infection necessitating treatment

Max Age: 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2011-09; Primary Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Total amount of sera withdrawn from the wound cavity | 4 weeks
  By each follow-up visit within the indicated time frame, the punctuated serum is collected and its volume is measured by a measuring cylinder acquired from the Pharmacy Department and data is recorded. At the end of the follow-up period, the total amount of serum (mL) is documented.

SECONDARY OUTCOMES:
Extent of early postoperative analgesic requirements | 4 days
  Assessment of analgesic consumption to achieve adequate pain relief for each patient. Pain relief is carried out according to institutional protocol and includes: diclofenac sodium, diclofenac sodium + orphenadrine, nalbuphine, metamizole sodium, paracetamole, tramadole.
Number of punctions following the removal of suction drain, and total volume of punctuated seroma (mL) | 4 weeks
Rate of local wound complications. | 4 weeks
Assessment of quality of life in the early postoperative period | 4 weeks
  Using EORTC QoL BR23, weekly for 4 weeks following surgery.
Mobility of the shoulder on the side of the operated side | 4 weeks
  Assessing shoulder motion on the 1st postoperative day, then weekly for 4 weeks.
  Abduction 1: 0°- 45° Abduction 2: 45° - 90° Abduction 3: 90° - 135° Abduction 4: 135° - 180°
Cost analysis | 4 weeks
  Suction drain, suction flask, syringes, number of patient-doctor consultations

CONTACTS AND LOCATIONS:
Overall Officials: Miklos Kasler, M.D., Ph.D., D.Sc., Prof., Principal Investigator — National Institute of Oncology; Laszlo Toth, M.D., Ph.D., Prof., Study Chair — National Institute of Oncology; Ferenc Renyi Vamos, M.D., Ph.D., Study Chair — National Institute of Oncology; Akos Savolt, M.D., Study Chair — National Institute of Oncology; Emil Farkas, M.D., Study Chair — National Institute of Oncology; Ildiko Horti, M.D., Study Chair — National Institute of Oncology; Zoltan Matrai, M.D., Principal Investigator — National Institute of Oncology
Locations (1):
- National Institute of Oncology, Budapest, Budapest, Hungary